CLINICAL TRIAL: NCT05548699
Title: PRO-MENTAL: Precision Mental Health in Diabetes - Subtypes of Mental Health, Trajectories, and Patterns With Glycaemic Control
Brief Title: Precision Mental Health in Diabetes - Subtypes of Mental Health, Trajectories, and Patterns With Glycaemic Control
Acronym: PRO-MENTAL
Status: Completed | Type: Observational
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Responsible Party: Principal Investigator, Norbert Hermanns, Prof. Dr. phil., Forschungsinstitut der Diabetes Akademie Mergentheim
Other Study IDs: HermannsNorbert2022-07-14VADM
Record Dates: First submitted 2022-09-09; First posted 2022-09-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus; Depressive Disorder; Depressive Symptoms; Anxiety Disorders; Anxiety and Fear; Eating Disorders; Eating Disorder Symptom; Eating Behavior; Hyperglycemia; Emotional Distress
MeSH Terms: conditions — Diabetes Mellitus; Depressive Disorder; Depression; Anxiety Disorders; Feeding and Eating Disorders; Feeding Behavior; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PRO-MENTAL is a non-interventional, prospective, observational study investigating longitudinal associations between diabetes distress, mental disorders, and glycemic outcomes in people with type 1 diabetes (T1D) and type 2 diabetes (T2D). The study aims to determine mental health subtypes, trajectories, and patterns and to advance a precision medicine approach to improve mental health in people with diabetes through personalized care and interventions.

A total of 1500 people with T1D or T2D will participate in the study, running over a 24-month period. Participants will be recruited at different levels of diabetes care including specialized centers and hospitals. The assessment includes a baseline assessment (clinical interview, questionnaire survey, and laboratory assessment) and four subsequent measurement time points - every six months - to a total period of two years. Each measurement time point includes an online questionnaire survey as well as a 14-day ambulatory assessment of daily mental and somatic variables (smartphone-based ecological momentary assessment (EMA) of daily sleep quality, mood, stress, and diabetes-related burdens/distress, as well as continuous glucose measurement (CGM) of daily glucose levels).

The study uses precision monitoring to identify evidence-based subgroups of people with diabetes with regard to mental disorders/problems and glycemic outcome. Epidemiological data regarding prevalence and incidence rates of depression, anxiety, and eating disorders will be analyzed, and patient trajectories and patterns will be determined. The study also aims to shed more light on the mediating mechanisms between mental health and glycemic outcomes.

The findings of the study will be used as the basis to develop a precision medicine approach with personalized interventions for specific sub-groups of people with type 1 and type 2 diabetes.

Note/Update 27.11.2025: The recruitment resulted in a total of 1290 participants enrolled until 31.12.2024 (= study completion date). Yet the recruitment and follow-up of participants is being continued within the ongoing TwinPeaks study (NCT07212075) from 2025-2027.

DETAILED DESCRIPTION:
Comorbid mental disorders as well as mental symptoms are common in people with type 1 diabetes (T1D) and type 2 diabetes (T2D). Depression, anxiety, and eating problems are particularly prevalent, and diabetes-related distress may contribute to or interact with mental disorders. Furthermore, while the management of diabetes aims to achieve near-normal glucose levels to prevent health decline and complications, glycemic outcomes may be impaired in people with significant mental comorbidity.

The objective of the PRO-MENTAL study is to use precision monitoring to identify evidence-based subgroups of people with diabetes with regard to mental disorders/problems and glycemic outcomes, to determine typical patterns and derive patient trajectories for informing a precision medicine approach offering personalized interventions for people with T1D and T2D. Precision monitoring uses continuous glucose monitoring (CGM) and ecological momentary assessment (EMA) methods as well as patient-reported outcomes (PRO) according to self-report scales and interviews.

Another aim is to answer epidemiological questions regarding depressive, anxiety and eating disorders in people with T1D and T2D (including assessment of bipolar disorders for differential diagnosis). In addition to clinical disorders, subclinical (=elevated) mental symptoms (e.g., depressive symptoms) and diabetes-related distress will be investigated as adverse factors in diabetes.

The findings of the study will serve as the basis for developing a precision medicine approach with personalized interventions for specific subgroups of people with T1D and T2D and mental comorbidity.

The primary research question refers to prospective associations of psychological disturbances/problems, especially depressive symptoms, anxiety symptoms, diabetes distress, and eating disorder symptoms, with self-management/health behaviors and glycemic outcomes. Using diagnostic interviews assessing affective, anxiety, and eating disorders and the collection of behavioral, somatic and psychological variables using questionnaires and surveys, subgroups and trajectories will be identified. In longitudinal analyses, the prognostic and moderating contribution of these parameters to the prediction of glycemic and mental health outcomes will be investigated.

Secondary objectives of the study are to identify predictors and/or moderators that may explain the incidence and persistence as well as associations between the above mental health variables and diabetes outcomes. For this purpose, measures of health-related quality of life, well-being, sleep quality, hypoglycemic anxiety, fear of sequelae, problems of diabetes treatment, diabetes acceptance, stressful life events, alcohol misuse, social support, COVID-19-related burden, and psychological resilience are also collected.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Diagnosis of type 1 diabetes (T1D) or type 2 diabetes (T2D)
* Diabetes duration ≥ 1 year
* Sufficient German language skills
* Written informed consent

Exclusion Criteria:

* Inability to consent,
* Significant cognitive impairment (e.g., cognitive disorder, dementia)
* Severe somatic disease or mental disorder likely to impede study participation or confound results (e.g., severe heart failure ≥ NYHA III; cancer requiring treatment; dialysis-dependent nephropathy; schizophrenia/psychotic disorder)
* Terminal illness
* Being bedridden

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Type 1 Diabetes or Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 1290 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of affective disorders at baseline (per diagnostic interview) | Baseline
  Diagnoses of affective disorders are assessed at baseline using the corresponding section of the Brief Diagnostic Interview for Mental Disorders (Mini-DIPS Open Access).
Prevalence of anxiety disorders at baseline (per diagnostic interview) | Baseline
  Diagnoses of anxiety disorders are assessed at baseline using the corresponding section of the Brief Diagnostic Interview for Mental Disorders (Mini-DIPS Open Access).
Prevalence of eating disorders at baseline (per diagnostic interview) | Baseline
  Diagnoses of eating disorders are assessed at baseline using the corresponding section of the Brief Diagnostic Interview for Mental Disorders (Mini-DIPS Open Access).
Depressive symptoms: incidence at 24-month FU | Baseline, 24-month FU
  Depressive symptoms are assessed with the Patient Health Questionnaire-9 (PHQ-9) at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU. Primary outcome is the incidence of depressive symptoms at 24-month FU compared to baseline.
Depressive symptoms: recovery at 24-month FU | Baseline, 24-month FU
  Depressive symptoms are assessed with the Patient Health Questionnaire-9 (PHQ-9) at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU. Primary outcome is the recovery from depressive symptoms at 24-month FU compared to baseline.
Anxiety symptoms: incidence at 24-month FU | Baseline, 24-month FU
  Anxiety symptoms are assessed with the Generalized Anxiety Disorders-7 (GAD-7) Questionnaire at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month. Primary outcome is the incidence of anxiety symptoms at 24-month FU compared to baseline.
Anxiety symptoms: recovery | Baseline, 24-month FU
  Anxiety symptoms are assessed with the Generalized Anxiety Disorders-7 (GAD-7) Questionnaire at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU. Primary outcome is the recovery from anxiety symptoms at 24-month FU compared to baseline.
Diabetes distress over time | Baseline, 24-month FU
  Diabetes distress is assessed with the Problem Areas in Diabetes Scale (PAID) at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU to detect changes in diabetes distress from baseline to 24-month FU.
Daily diabetes burdens over time | Baseline, 24-month FU
  Daily diabetes burdens (daily diabetes distress) are assessed at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU over each 14 consecutive days using smartphone-based ecological momentary assessment with selected items of the Problem Areas in Diabetes Scale (PAID) adapted for daily assessment (rated on an 11-point scale from 0 - 10) to detect changes in daily burdens from baseline to 24-month FU.
Eating problems: incidence | Baseline, 24-month FU
  Eating problems (=disordered eating behavior/eating disorder symptoms) are assessed with the Diabetes Eating Problems Survey-Revised (DEPS-R; a validated, self-report measure for eating problems of people with diabetes where generic eating disorder questionnaires yield significant false-positive rates due to specific eating behaviors and dietary requirements for diabetes) at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU. Primary outcome is the incidence of eating problems at 24-month FU compared to baseline.
Glycated hemoglobin (HbA1c) over time | Baseline, 24-month FU
  HbA1c (glycated hemoglobin), a laboratory measure of average blood glucose over the past 8 to 12 weeks, is estimated/collected at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU from the participants to detect changes for glycated hemoglobin from baseline to 24-month FU.
Glycemic levels (CGM glucose) over time | Baseline, 24-month FU
  In addition to the global parameter HbA1c, automatically recorded daily glucose values are obtained from participants where continuous glucose monitoring (CGM) devices are used. Available glucose data are extracted at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU for each over 14 consecutive days of CGM measurement - parallel to the daily EMA - to detect changes in glucose levels from baseline to 24-month FU.
Daily stress levels over time | Baseline, 24-month FU
  Daily stress levels are assessed at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU over each 14 consecutive days using smartphone-based ecological momentary assessment with items from the previous DIA-LINK study (requesting the current stress level and specific stressors, rated on an 11-point scale from 0 - 10) to detect changes in daily stress levels from baseline to 24-month FU.

SECONDARY OUTCOMES:
General health state over time | Baseline, 24-month FU
  The self-evaluated general self-rated health state is assessed at baseline, 12-month FU, and 24-month FU using the 8-item Short Form Health Survey (SF-8) to detect changes in the health state from baseline to 24-month FU.
Subjective health over time | Baseline, 24-month FU
  The subjective health state is assessed at baseline, 12-month FU, and 24-month FU using the visual analogue scale (VAS) of the EuroQol Five Dimensions Questionnaire (EQ-5D) to detect changes in subjective health from baseline to 24-month FU.
Wellbeing over time | Baseline, 24-month FU
  Wellbeing is assessed at baseline, 12-month FU, and 24-month FU using the WHO-Five Well-being Index (WHO-5) to detect changes in wellbeing from baseline to 24-month FU.
General sleep quality over time | Baseline, 24-month FU
  General sleep quality assessed at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU using items of the Pittsburgh Sleep Quality Index (PSQI) to detect changes in sleep quality from baseline to 24-month FU.
Daily sleep quality over time | Baseline, 24-month FU
  Daily sleep quality assessed at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU over each 14 days using smartphone-based ecological momentary assessment with selected PSQI items adapted for daily assessment (rated on an 11-point scale from 0 - 10) to detect changes in daily sleep quality from baseline to 24-month FU.
Fear of diabetes complications over time | Baseline, 24-month FU
  Fear of diabetes complications is assessed at baseline, 12-month FU, and 24-month FU with the short form of the Fear of Diabetes Complications Questionnaire (FDCQ; requesting frequencies of worries and fears regarding long-term complications of diabetes) to detect changes in fear levels from baseline to 24-month FU.
Fear of hypoglycemia over time | Baseline, 24-month FU
  Fear of hypoglycemia is assessed at baseline, 12-month FU, and 24-month FU with the short form of the Hypoglycemia Fear Survey II (HFS-II-SF; requesting hypoglycemia-related worries and avoidance behaviors) to detect changes in fear levels from baseline to 24-month FU.
Diabetes acceptance over time | Baseline, 24-month FU
  Diabetes acceptance is assessed at baseline, 12-month FU, and 24-month FU with a short form of the Diabetes Acceptance Scale (DAS) to detect changes in diabetes acceptance from baseline to 24-month FU.
Daily eating problems over time | Baseline, 24-month FU
  Eating problems in daily life are assessed at baseline, 6-month FU, 12-month FU, 18-month FU, and 24-month FU over each 14 consecutive days using smartphone-based ecological momentary assessment with items requesting specific problematic eating behaviors (rated on an 11-point scale from 0 - 10) to detect changes in daily eating problems from baseline to 24-month FU.
Diabetes self-management over time | Baseline, 24-month FU
  Diabetes self-management behaviors are assessed at baseline, 12-month FU, and 24-month FU with the revised Diabetes Self-Management Questionnaire-Revised (DSMQ-R) to detect changes in diabetes self-management from baseline to 24-month FU.
Alcohol misuse over time | Baseline, 24-month FU
  Alcohol abuse/misuse is assessed at baseline, 12-month FU, and 24-month FU using the 5-item alcohol module of the Patient Health Questionnaire (PHQ-D) to detect changes in alcohol use from baseline to 24-month FU.

OTHER OUTCOMES:
COVID-19-related burden | Baseline, 24-month FU
  COVID-19-related burden is assessed as control variable at baseline, 12-month FU, and 24-month FU with items from the previous DIA-LINK studies requesting the burden due to the pandemic (rated on an 11-point scale from 0 - 10).
Psychological resilience | Baseline
  Psychological resilience is assessed as control variable at baseline with the 13-item Resilience Scale (RS-13).
Social support | Baseline, 24-month FU
  Social support is assessed as control variable at baseline, 12-month FU, and 24-month FU with the 3-item Oslo Social Support Scale (OSSS-3).
Night eating | Baseline, 24-month FU
  Night eating behaviors are assessed as control variable at baseline, 12-month FU, and 24-month FU with the Night Eating Questionnaire (NEQ).
Stressful life events | Baseline, 24-month FU
  Stressful life events during the past 12 months are assessed as control variable at baseline, 12-month FU, and 24-month FU using the Life Events Questionnaire (LEQ) (=the German "Fragebogen zu kritischen Lebensereignissen"; reflecting the overall burden due to stressful life events in the past year).

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Hermanns, Prof, PhD, Principal Investigator — Research Institute Diabetes Academy Mergentheim (FIDAM); Bernhard Kulzer, Prof, PhD, Principal Investigator — Research Institute Diabetes Academy Mergentheim (FIDAM)
Locations (2):
- Germany (2):
  - Diabetes Center Mergentheim, Bad Mergentheim, Baden-Wurttemberg
  - Diabetes Practice Mergentheim, Bad Mergentheim, Baden-Wurttemberg

REFERENCES:
- See also: ClinicalTrials entry of the "TwinPeaks" study that has continued the recruitment and follow-up of the PRO-MENTAL cohort since 2025. — https://clinicaltrials.gov/study/NCT07212075